CLINICAL TRIAL: NCT00467181
Title: A Pilot Study to Investigate Fenoldopam Usage in the Prevention of Postoperative Renal Dysfunction in Patients at a High Risk for Renal Impairment During Cariopulmonary Bypass for Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Dr. William Fallon, Summa Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP05009
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2007-04

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass
Keywords: cardiac surgery; renal dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — Fenoldopam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fenoldopam

SUMMARY:
The Primary objective is to reduce the incidence of postoperative renal dysfunction in a high-risk subset of patients undergoing cardiac surgery on cardiopulmonary bypass with Fenolopam, a selective dopamine-1 receptor agonist. Perioperative renal function will be observed in 3 randomly selected groups of patients-Fenoldopam infusion at 0.03 cg/kg/min, Fenoldopam at 0.1 mcg/kg/min or placebo

Secondary objective: will be to correlate Fenoldopam usage with postoperative clinical outcomes such as ICU stay, hospital stay, need for inotropes/vasopressors, need for diuretics, requirements for ECF at discharge, and overall perioperative cost reduction through decreased ICU and hospital length of stay.

DETAILED DESCRIPTION:
Although all patients undergoing cardiac surgery are at risk for renal dysfunction, there are certain preoperative clinical parameters which have been shown to place patients at particularly high risk for postoperative renal demise. These factors include age greater than 70 (with those patients greater than 80 years being at particular high risk), history of New York Heart Association Class 3 or 4 congestive heart failure, previous coronary artery bypass grafting, pre-operative creatinine level 1.24-1.77 mmol/dL, type I diabetes, preoperative glucose >166 mmol/dL, cardiopulmonary bypass time >3 hours, and low cardiac output states (those states requiring intra-aortic balloon pump (IABP) or with cardiac index of less than 1.5 or requiring more than 3 inotropic drugs).1 Recently, there has been interest in the pharmacologic manipulation of peripheral dopamine receptors (DA1 and DA2) in an attempt to augment and preserve renal function. Goldberg and colleagues localized DA1 receptors to vascular smooth muscle postsynaptic membranes in renal, coronary, cerebral, mesenteric, and peripheral artery vasculature, in the proximal convoluted tubule, and in the cortical collecting ducts of the nephron.6,7 Stimulation of the DA1 receptor activates adenylate cyclase causing vascular smooth muscle vasodilation and naturesis with increased urinary sodium excretion by inhibiting sodium-potassium ATPase-dependent processes at the proximal convoluted tubule and the thick portion of the ascending loop of Henle.6,8,9 The greatest effect of DA1 receptor activation occurs in the renal vasculature (mostly at afferent arteriole)9, causing an increase of renal blood flow up to 35% in normal patients and up to 77% in those patients with renal vascular disease.10,11 DA2 receptors are found in the renal parenchyma, presynaptic nerve terminals of adrenergic nerves and sympathetic ganglia, and in the adrenal cortex.10 DA2 receptor activation leads to inhibition of norepinephrine release (as part of a negative feedback loop) and inhibition of angiotensin II mediated release of aldosterone.10,12 With activation of DA2 receptors in the kidney, a resultant decrease in renal blood flow, decrease in glomerular filtration rate, and decrease in diuresis and naturesis is observed, effects that are opposite to and may offset DA-1 receptor agonism. Mayes and colleagues showed no improvement in renal function in patient undergoing CABG with "renal-dose" dopamine.6, 13 It is theorized that dopamine's inability to provide renal protection may be due to its lack of specificity for DA-1 receptors and resultant dose-dependent agonism for DA-2 receptors and alpha1-adrenergic receptors.6, 14, 15 As mentioned, dopamine's activation of these receptors results in decreased renal blood flow, glomerular filtration rate, and sodium excretion6, 16, thereby offsetting the effects of DA-1 receptor agonism.

Fenoldopam is the first commercially available selective DA1 receptor agonist. Fenoldopam is a selective agonist for DA1 receptors with no activity at DA2 receptors, alpha adrenergic receptors, or beta adrenergic receptors. Currently, Fenoldopam is used as an intravenous infusion for hypertensive emergencies. When given to hypertensive patients in doses of 0.025-0.5 mcg/kg/min, a reduction in blood pressure is seen in a linear and dose dependent manner.9, 17, 18, 19, 20 Despite reductions in perfusion pressure, glomerular filtration rate and renal blood flow are equivalent or even increased.9, 20, 21 When given to normotensive patients at doses of 0.03-0.3 mcg/kg/min, Vandana and colleagues have shown that Fenoldopam significantly increased renal blood flow in a dose-dependent manner when compared with placebo with no change in systolic blood pressure and minimal changes in diastolic blood pressure (1 mmHg @ 0.3 mcg/kg/min dose) and heart rate (14 bpm @ 0.3 mcg/kg/min dose). In addition, there were no serious or severe side effects even at the highest doses.9 These observations are consistent with prior studies of Fenoldopam in both normotensive22 and hypotensive23 patients. Fenoldopam's lack of effects on venous capacitance as well as the lesser role that resistance plays in determining blood pressure in normotensive patients may further explain the negligible effect that Fenoldopam has on blood pressure in normotensive subjects. This leads to a theoretic "renal protection" provided by Fenoldopam at doses which elicit negligible deleterious effects.

As mentioned, Fenoldopam is a selective DA1 receptor agonist created through modification of the dopamine molecule with the addition of chloride, sulfur, and a benzene ring.10 These changes result in agonistic effects exclusively on the DA-1 receptor with no DA2 receptor activation and no direct or indirect actions on both alpha and beta adrenergic receptors.10 Fenoldopam has a short half-life of 5-10 minutes, a linear relationship between plasma concentration and infusion rate, and a small volume of distribution allowing rapid intravenous titration.24 These characteristics make Fenoldopam ideal for intravenous infusion with a steady-state plasma concentration being achieved within 30-60 minutes, steady-state concentrations remaining constant during infusion, and with a negligible concentration (<0.2 mcg/L) 2 hours after discontinuation as demonstrated by Allison and colleagues.24 Hepatic clearance of Fenoldopam occurs through conjugation via sulfation or glucuronidation.10 Klecker and colleagues demonstrated that drug-drug interactions are negligible due to parallel pathways of metabolism.25 Recent studies by Garwood and colleagues and Caimmi and colleagues have shown preservation of renal function by perioperative infusion of Fenoldopam as indicated by lower creatinine level at discharge in those patients at high risk for perioperative renal demise.26, 27 However, a prospective randomized control trial has yet to be performed. There is also uncertainty that these reductions in serum creatinine levels at discharge are of any practical benefit in terms of reduced morbidity, reduced length of stay, reduced cost, or improved clinical performance. In addition, an optimal dose for Fenoldopam for this clinical indication has yet to be determined. For this pilot study, Fenoldopam will be infused at 0.03 mcg/kg/min or 0.1 mcg/kg/min. These doses were chosen due to their proven effectiveness to significantly increase renal blood flow with minimal effects on blood pressure and heart rate.9 The goal of this study is to evaluate the effectiveness of Fenoldopam, a new selective dopamine-1 receptor agonist, in the reduction of postoperative renal dysfunction in a high-risk subset of patients undergoing cardiac surgery in a prospective randomized control pilot study. This will be accomplished through infusion of Fenoldopam at 0.03 mcg/kg/min, 0.1 mcg/kg/min, or placebo in a double blinded, randomized, prospective trial where postoperative creatinine, urine output, and progression to renal dysfunction will be observed. Renal dysfunction will be defined as an increase in serum creatinine by greater than 50% of the preoperative value or a serum creatinine that exceeds 2.0 mg/dL at any time postoperatively prior to discharge.. In addition, length of ICU stay, length of hospital stay, ventilator requirements, need for diuretics, need for perioperative inotropes/vasopressors, and need for discharge to extended care facilities will be examined for each group. The null hypothesis is that Fenoldopam will not reduce the incidence of postoperative renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing CABG, CABG/valve operations must meet one of the following:

* Age greater than 70
* Preoperative (within one week) creatinine > or = 1.3
* Insulin depenent diabetes
* NYHA CHF class 3 or 4
* Bypass time anticipated to be greater than 3 hours
* Redo coronary artery bypass grafting
* Low cardiac output states -need for inotropic agents or IABP preoperatively

Exclusion Criteria:

* Emergent operations
* Preopertive liver failure
* Preopertive acute or chronic dialysis dependence
* Known allergy to Fenoldopam
* Patients in whom usage of dopaminergic medications are contraindicated
* Age less than 30
* Caridac surgery without cardiopulmonary bypass
* Patients acively participating in other clinical trials
* Usage of dopaminergic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To evaluate postop renal dysfunction in patients undergoing cardiac surgery. Post-op creatinine, urine output, and progression to renal dysfunction will be observed. Renal dysfunction will be defined as an increase in | During Stay

SECONDARY OUTCOMES:
Length of ICU and hospital stay, ventilator requirements,need for diuretics, or perioperative inotropes/vasopressors, and need for discharge to extended care facilities. | Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Marion Hochstetler, MD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014